CLINICAL TRIAL: NCT02182687
Title: A Randomized Phase II Study of Individualized Stereotactic Body Radiation Therapy (SBRT) Versus Trans-Arterial Chemoembolization (TACE) With DEBDOX Beads as a Bridge to Transplant in Hepatocellular Carcinoma.
Brief Title: Stereotactic Body Radiation Therapy (SBRT) Versus Trans-Arterial Chemoembolization (TACE) as Bridge to Liver Transplant
Acronym: SBRTvsTACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCID 2014-026
Record Dates: First submitted 2014-06-23; First posted 2014-07-08 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; HCC
Keywords: Hepatocellular carcinoma (HCC); Orthotopic liver transplant; Bridge to transplant; stereotactic body radiation therapy (SBRT); trans-arterial chemoembolization (TACE)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiotherapy; Chemoembolization, Therapeutic; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Other): Stereotactic Body Radiation Therapy (SBRT)
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Arm B (Other): Trans-Arterial Chemoembolization (TACE) Drug: Doxorubin
  Interventions: Procedure: Trans-Arterial Chemoembolization (TACE); Drug: Doxorubin

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered in five total fractions, with at a minimum of one day between any two treatments. The entire treatment must be delivered within 15 total days.
  Other Names: Radiation Therapy
  Arms: Arm A
Procedure: Trans-Arterial Chemoembolization (TACE) — First day will be administered and a second TACE will be administered after 4 weeks and subsequently if imaging is showing disease progression. Following each TACE procedure all patients will remain in hospital for observation.
  Other Names: Chemoembolization
  Arms: Arm B
Drug: Doxorubin — This procedure will be completed with 2 vials of drug eluting beads each loaded with 50 mg of Doxorubin.
  Other Names: Doxorubin bead therapy
  Arms: Arm B

SUMMARY:
This study will compare stereotactic body radiation therapy (SBRT) to trans-arterial chemoembolization (TACE) as a bridging strategy for patients with HCC undergoing orthotopic liver transplantation. We propose that SBRT will be associated with longer time intervals between initial treatment and the need for retreatment, compared to TACE, as a "bridge" to orthotopic liver transplantation.

DETAILED DESCRIPTION:
For patients with hepatocellular carcinoma (HCC) who are waiting for a liver transplant, local treatment of their disease has become the standard of care in an effort to decrease dropout rates and as a means of reducing tumor recurrence after transplantation. However, the best modality for patients undergoing treatment as a bridge to transplantation is unclear. This study will compare stereotactic body radiation therapy (SBRT) to trans-arterial chemoembolization (TACE) as a bridging strategy for patients with HCC undergoing orthotopic liver transplantation. We propose that SBRT will be associated with longer time intervals between initial treatment and the need for retreatment, compared to TACE, as a "bridge" to orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria

* Patients with hepatocellular carcinoma are eligible for this trial.

Hepatocellular carcinoma is defined as having at least one of the following:

Biopsy proven hepatocellular carcinoma (HCC); or A discrete hepatic tumor(s) as defined by the Barcelona (29) criteria for cirrhotic patients, >2cm with arterial hypervascularity and venous or delayed phase washout on CT or MRI.

* Patient is within Milan Criteria and "listed" for orthotopic liver transplantation.
* Patients must have a Zubrod performance status of ≤2.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must be 18 years of age or older. Adult patients of all ages, both sexes and all races will be included in this study.
* Patients must be Child-Turcotte-Pugh (CTP) Class A or Class B (≤ 7).
* Female patients within reproductive years may not be, nor become, pregnant during participation in this study. Both male and female patients within reproductive years must agree to use an effective contraceptive method during treatment. Women of childbearing age will be required to undergo a urine or serum pregnancy test to ensure they are not pregnant.
* Patients must have adequate organ function within 2 weeks of enrollment. Bone marrow: Platelets ≥30,000/mm3 Renal: BUN ≤40 mg/dl; creatinine ≤2.0 mg/dl Hepatic: INR ≤ 1.5 or correctable by Vitamin K, unless anti- coagulated for another medical reason Bilirubin < 3 mg/dl (in the absence of obstruction or pre-existing disease of the biliary tract, e.g. primary sclerosing cholangitis) Patients uninvolved liver volume will be estimated and must be > 700ml.
* Patients must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the Lahey Hospital and Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.

Exclusion Criteria

* Patients in a "special category" designated the Public Health Service, including patients younger than 18, pregnant women, and prisoners.
* Refractory ascites or ascites that requires paracentesis for management.
* Patients with a solitary lesion greater than 5.0cm in size or more than 2 discrete lesions the largest greater than 3.0 cm in size.
* Known allergy to intravenous iodinated contrast agents unresponsive to prednisone pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Nugent, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 24 | 30
Completed | 19 | 29
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 60 pts were consented, 12 pts failed to undergo treatment. Among the 12 not treated, 6 pts were screen failures. Additionally, 4 pts were randomized but declared ineligible before treatment. Two more pts underwent treatment and were excluded from analysis: 1 pt treated on the SBRT arm was misdiagnosed (large cell lymphoma) and 1 pt on the TACE arm was lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 19 | 29 | 48
Age, Continuous [Median (Standard Deviation); unit: years] | 63.2 (4.6) | 61.7 (6.2) | 62.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 16 | 23 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 29 | 48

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Progression Over Time
Description: Time from SBRT and TACE intervention to progression was tracked for subject receiving protocol intervention. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion.
Time Frame: 3, 6 and 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of patients with progression
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 29
percentage of patients with progression
  3 Month | 0 [0 to 0] | 3.4 [0.5 to 22.1]
  6 Month | 0 [0 to 0] | 26.5 [13.5 to 47.9]
  12 Month | 11.1 [1.6 to 56.7] | 38.0 [21.1 to 61.8]

2. Secondary Outcome: Toxicity To Compare Participants With Treatment-related Adverse Events as Assessed by CTCAE
Description: Grade 3 or greater toxicity with treatment-related adverse events was tracked at protocol specific time points. Grading of events was according to CTCAE.
Time Frame: At each treatment, 2 weeks post treatment, 2 months post treatment, 5 months post treatment, every 3 months until 24 months post treatment
Population: Subjects in both arms were observed for adverse events at protocol specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 29
Participants | 1 | 3

3. Secondary Outcome: Number of Participants Who Require Further Interventions Prior to Liver Transplant
Description: Each patient on each arm was followed to see how if further treatment interventions were needed prior to liver transplant. This outcome summarizes the number of participants who needed further treatment.
Time Frame: 2 weeks post treatment, 2 months post treatment, 5 months post treatment, every 3 months until 24 months post treatment
Measure: Number; unit: participants
Groups:
- Arm A SBRT: ARM A is patients randomized to SBRT.
- TACE Arm B: TACE
Arm/Group | Arm A SBRT | TACE Arm B
Number analyzed (Participants) | 19 | 29
participants | 1 | 6

4. Secondary Outcome: Pathologic Response of Treated Lesion(s)
Description: Pathologic complete response was recorded for patients in both arms after completion of liver transplant. Explanted liver was reviewed by the pathologist to determine if residual tumor was identified.
Time Frame: At time of liver transplant
Population: Patients undergoing liver transplant were reviewed for complete pathologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 29
Participants
  Count of participants undergoing Liver Transplant | 15 | 20
  Patients having a complete pathologic response to therapy | 4 | 7
  Patients having additional HCC outside the treated area | 6 | 8

5. Secondary Outcome: Radiologic Response of Treat Lesion(s)
Description: Number of patients with a radiographical response to treatment.The status of each treated tumor/target lesion was assessed by MRI or CT scan and classified as progression if there was tumor growth (excluding growth due to biloma or abscess formation), residual or new enhancement of the ablated tumor (excluding benign peri-ablational enhancement), or contiguous viable tumor as determined by mRECIST Criteria.
Time Frame: Baseline, 3 months post-treatment, 6 months post-treatment, every 3 months thereafter until 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 29
Participants | 18 | 23

6. Secondary Outcome: Quality of Life - Questionnaires Include PIQ-6 and SF-36v2 Health Survey
Description: Quality of life was assessed with Short Form 36 Health Survey (SF-36v2®) and Pain Impact Questionnaire (PIQ-6TM) Health Survey. Data was stored and scored with Pro CoRE 2.0 Smart Measurement® System. Scores were analyzed at three time points, baseline-before the first treatment, acute response-2 weeks post the first treatment, and long term response - 6 months after the first treatment.
  The PIQ-6 Pain Impact Questionnaire measures how a subject's pain affects every day activities. The SF-36v2 Health Survey measures functional health and well-being from the subject's point of view. The survey's scores range from 0-100, with 0 having the most disability and a score of 100 being equivalent to no disability.
Time Frame: Baseline, 2 weeks post-treatment, 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 29
score on a scale
  SF36-Mental Component Score (baseline) | 50.2 (9.4) | 49.9 (7.6)
  SF36-Mental Component Score (2-week) | 49.7 (9.8) | 48.7 (8.8)
  SF36-Mental Component Score (6 Months) | 53.8 (7.1) | 50.9 (8.3)
  SF36-Physical Component Score (baseline) | 48.1 (9.7) | 48.3 (9.0)
  SF36-Physical Component Score (2 weeks) | 44.2 (9.8) | 44.7 (9.5)
  SF36-Physical Component Score (6 Months) | 49.6 (5.8) | 45.1 (10.3)
  Pain Summary score -hand weighted (baseline) | 49.9 (9.3) | 49.5 (10.0)
  Pain Summary Score - hand weighted (2 weeks) | 51.4 (8.0) | 54.2 (9.8)
  Pain Summary Score - hand weighted (6 Months) | 47.2 (8.3) | 50.1 (8.7)

ADVERSE EVENTS:
Time Frame: Baseline, During Treatment, post treatment follow-up visit, 3 Month, 6 Month, then every 3 months until 24 month time point.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/19 | 1/29
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/29
Other Adverse Events (participants affected / at risk) | 7/19 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=29)
Gastritis and GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
biliary infection (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=29)
RILD with refractory ascities (Hepatobiliary disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 6 (6) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
bacterial peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
WBC decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
hypertension (Vascular disorders) | 1 (1) | 4 (4)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
hepatic infarct (Hepatobiliary disorders) | 0 (0) | 1 (1)
esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
One primary limitation was the small, single institution, randomized phase II design. Given the small overall numbers, no definitive judgements can be made.

Another potential weakness of the trial was the selection of our primary endpoint. Our primary endpoint was time to residual or progressive cancer in the previously treated lesion(s).

A third limitation of this trial was incomplete compliance with QOL questionnaires. Lastly, our QOL measures were performed over a long interval.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT02182687/Prot_SAP_000.pdf